CLINICAL TRIAL: NCT00805532
Title: Behavioral Activation for PTSD, Depression Treatment in OIF/OEF Veterans
Brief Title: Behavioral Activation for PTSD/Depression Treatment in OIF/OEF Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-019-06F; PVAMC ID: 1738 (Other: PVAMC R&D); VA PSHCS SUB IRB ID: 33950 (Other: VA PSHCS R&D); Grant #: 08-0306 (Other Grant/Funding Number: VA Clinical Science R&D)
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-04

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: PTSD; depression; behavior therapy; veterans; behavioral activation; usual care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation (Experimental): Behavioral Activation (BA), modified to be delivered in 6-8, 60 minute sessions to address PTSD-related problems.
  Interventions: Behavioral: Behavioral Activation treatment
- Treatment as Usual (Active Comparator): Treatment As Usual for PTSD (TAU) within VA PTSD specialty clinics. Actual clinical practice varies between sites and between providers within sites, as is typical of the VA health care system.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Behavioral Activation treatment — Behavioral Activation (BA) is a present-focused psychotherapy based on behavioral theory and principles of change, that aims to re-engage individuals with meaningful and pleasurable life activities by targeting and problem-solving patterns of avoidance. It is well-established as a treatment for depression and has been modified for the current study to address PTSD-related problems.
  Other Names: BA
  Arms: Behavioral Activation
Other: Treatment as Usual — Usual Care for PTSD (UC)-that is provided in the VA PTSD Specialty clinics. Actual clinical practice varies between sites and between providers within sites, as is typical of the VA health care system. Subjects assigned to Usual Care will be permitted to receive medical intervention (i.e., pharmacotherapy) and any additional psychotherapy deemed appropriate by the provider. They will also be offered a minimum of 6 sessions of individual therapy.
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
The present study is a randomized, controlled trial that compares Behavioral Activation (BA) to Treatment As Usual (TAU) in PTSD Specialty clinics, as early psychotherapeutic interventions for OIF/OEF veterans with posttraumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
A sizable proportion of soldiers involved in the Iraq and Afghanistan conflicts are experiencing mental health and adjustment problems on their return, including posttraumatic stress disorder and depression (Hoge et al., 2004). Both PTSD and depression can be chronic and debilitating disorders, associated with impairments in social, occupational, and physical functioning, as well as high health care utilization (Katon, Unutzer, & Simon, 2004; Stein et al., 2005).

Although empirically supported treatments exist for established PTSD and depression, much less is known about effective early interventions for these conditions. Exploration of early intervention options is necessary, particularly in the case of the new veteran population, as such interventions could address social, occupational and physical impairments before they become too intractable. Also, successful early interventions could curtail high health care utilization dramatically across time. The development of such early interventions for PTSD and depression must also take into account any specifications of accessibility and acceptability that are particular to the OIF/OEF veteran population.

The present study is a randomized, controlled trial that compares Behavioral Activation (BA), to Treatment As Usual (TAU) as early interventions for OIF/OEF veterans with posttraumatic stress disorder (PTSD). Participants will be recruited largely from the primary health care setting (to increase acceptability and accessibility to the veteran population). Both BA and TAU treatment groups will be administered by psychotherapists who specialize in the treatment of PTSD. Both groups will be assessed at pre-, mid- and post-treatment time points to determine change over time, health care utilization and treatment satisfaction. This is a dual-site study that will be carried out at both the Portland VA Medical Center (PVAMC) and the VA Puget Sound Health Care Center (VA PSHCS) and coordinated at the PVAMC.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with assessment and therapy schedule.
* Ability to comply with study regulations.
* English fluency.
* Must meet diagnostic criteria for PTSD (related to trauma experienced during military service). PTSD will be assessed using the Clinician-Administered PTSD Scale for DSM-IV (CAPS; Blake, Weathers, Nagy, Kaloupek, Charney & Keane, 2003).

Exclusion Criteria:

* Bipolar disorder.
* Psychotic disorders.
* Substance dependence. Because these conditions warrant alternative treatments. Bipolar, psychotic and substance dependence disorders will be assessed using the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I; First, Spitzer, Gibbon & Williams, 2002).
* Report active and imminent suicidal intent. If imminent suicidality is present, this would suggest that a treatment specifically targeting this intent is indicated. Suicidal intent will be assessed using The Brief Assessment for Suicidal Ideation or Behavior that was designed for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy W. Wagner, PhD, Principal Investigator — VA Medical Center, Portland
Locations (2):
- United States (2):
  - VA Medical Center, Portland, Portland, Oregon
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in the publications
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 6 months after publication of the manuscript(s)
Access Criteria: The PIs will review requests and consult with the R&D offices and privacy officers at both sites prior to release of data.

REFERENCES:
- [Derived] Wagner AW, Jakupcak M, Kowalski HM, Bittinger JN, Golshan S. Behavioral Activation as a Treatment for Posttraumatic Stress Disorder Among Returning Veterans: A Randomized Trial. Psychiatr Serv. 2019 Oct 1;70(10):867-873. doi: 10.1176/appi.ps.201800572. Epub 2019 Jul 24. PMID 31337325

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Activation (BA): Behavioral Activation (BA)-BA is a present-focused, well-established treatment for depression that targets patterns of avoidance and involves the identification and enactment of activities that are reinforcing to the individual and consistent with his/her long-term goals. BA has been modified to address PTSD concerns in addition to depression and to be delivered in 6-8, 60-minute sessions. It was delivered by skilled psychotherapists.
- Treatment as Usual (TAU): Participants randomized to Treatment as Usual (TAU) were referred for treatment within the PTSD Clinical Teams at the VAPORHCS and PSHCS. In both clinics providers are trained in Prolonged Exposure therapy (PE) and Cognitive Processing Therapy (CPT). Both clinics also offer skills-based "coping skills" treatments for PTSD and pharmacotherapy. Actual treatment received was determined collaboratively between the PTSD Clinic Care provider and veteran and could include any of these treatment options or combinations of treatments.
Period: Overall Study
Arm/Group | Behavioral Activation (BA) | Treatment as Usual (TAU)
Started | 42 | 39
Completed | 42 (We did intent-to-treat analyses so 42 participants' data were analyzed.) | 38
Not Completed | 0 | 1
Not completed — invalid data | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation (BA) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (6.4) | 30.0 (7.1) | 30.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 39 | 36 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska Native | 0 | 1 | 1
  Race/Ethnicity: Asian or Native Hawaiian or Pacific Islander | 2 | 2 | 4
  Race/Ethnicity: Black or African American | 2 | 2 | 4
  Race/Ethnicity: White Not Hispanic | 34 | 28 | 62
  Race/Ethnicity: White Hispanic | 1 | 2 | 3
  Race/Ethnicity: Other | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 42 | 38 | 80

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS-IV)
Description: The CAPS is a clinician-administered scale and is considered the "gold standard" for assessing the presence of PTSD. Items are ranked on Likert scales according to both frequency (0=never to 4=daily or almost every day) and intensity (0=none to 4=extreme) of symptoms, yielding an overall severity score by summing frequency and intensity ratings (range 0 to 136, with higher scores reflecting greater symptomatology). Scale scores corresponding to the 3 subcategories of PTSD symptoms (intrusive symptoms, avoidance symptoms, and hyperarousal symptoms) can be similarly obtained (scores range from 0-40, 0-56, 0-40 for the 3 subscales, respectively). Internal consistency, interrater reliability, and validity of this measure are strong and well-documented.
Time Frame: Pre-treatment, post-treatment (12 weeks after 1st therapy session), and 3-month follow-up (24 weeks after first therapy session)
Population: OIF/OEF Veterans with PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Behavioral Activation: Behavioral Activation (BA)- modified to be delivered in 6-8, 60 minute sessions in to address PTSD-related problems.
  Behavioral Activation treatment: Behavioral Activation (BA) is a present-focused psychotherapy based on behavioral theory and principles of change, that aims to re-engage individuals with meaningful and pleasurable life activities by targeting and problem-solving patterns of avoidance. It is well-established as a treatment for depression and has been modified for the current study to address PTSD-related problems.
- Treatment as Usual: Treatment As Usual for PTSD (TAU)-that is provided in the VA PTSD Specialty clinics. Actual clinical practice varies between sites and between providers within sites, as is typical of the VA health care system. Subjects assigned to TAU will be permitted to receive medical intervention (i.e., pharmacotherapy) and any additional psychotherapy deemed appropriate by the provider. They will also be offered a minimum of 6 sessions of individual therapy.
  Treatment as Usual: Usual Care for PTSD (UC)-that is provided in the VA PTSD Specialty clinics. Actual clinical practice varies between sites and between providers within sites, as is typical of the VA health care system. Subjects assigned to Usual Care will be permitted to receive medical intervention (i.e., pharmacotherapy) and any additional psychotherapy deemed appropriate by the provider. They will also be offered a minimum of 6 sessions of individual therapy.
Arm/Group | Behavioral Activation | Treatment as Usual
Number analyzed (Participants) | 42 | 38
units on a scale
  Pre Treatment | 75.9 (15.2) | 82.0 (15.7)
  Post Treatment | 54.4 (23.0) | 70.1 (25.7)
  3-Mo Follow-Up | 56.25 (25.4) | 64.6 (28.3)

2. Secondary Outcome: Posttraumatic Stress Disorder Checklist-Military Version (PCL-M)
Description: The PCL-M is a 17 item self-report scale that assesses the presence of DSM-IV PTSD symptoms. Items are rated on a 5-point Likert scale (1= not at all to 5=extremely) according to how much the symptom bothered the respondent over the past month. Scores range from 17-85 with higher scores representing greater symptom severity.
Time Frame: Pre-treatment, post-treatment (12 weeks after first therapy appointment), 3-month follow-up (24 weeks after first therapy appointment)
Population: OIF/OEF Veterans with PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) | Treatment as Usual (TAU)
Number analyzed (Participants) | 42 | 38
units on a scale
  Pre-Treatment | 59.0 (7.7) | 59.0 (8.1)
  Post-Treatment | 44.1 (12.0) | 52.6 (13.0)
  3-Mo Follow-Up | 48.0 (13.4) | 51.4 (15.1)

3. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The Beck Depression Inventory-II (BDI-II) (Beck, Steer, & Brown, 1996) is a 21-item measure of subjective levels of depression. Items are rated on Likert-scales from 0-3 (individual descriptions are provided for each number ranging from the absence of the symptom to the severe manifestation of the symptom). Scores can range from 0-63 with higher scores representing higher levels of depression. This widely used measure of depression is commonly included in outcome studies in order to determine treatment effects on severity of depressive symptoms and has excellent psychometric properties.
Time Frame: as for outcome 2
Population: OIF/OEF Veterans with PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) | Treatment as Usual (TAU)
Number analyzed (Participants) | 42 | 38
units on a scale
  Pre-Treatment | 24.8 (7.0) | 25.2 (8.2)
  Post-Treatment | 17.5 (10.4) | 23.3 (11.4)
  3-Mo Follow-Up | 21.0 (10.0) | 21.5 (11.8)

4. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: The Sheehan Disability Scale (SDS) (Sheehan, 2000) is a three item self-rated scale of impairment that is widely used in psychopharmacology studies (allowing comparison with these studies). The items ask the respondent to rate (on a Likert scale of 0-10, unimpaired to highly impaired) to what extent their symptoms interfere with their functioning in the areas of: work, social, and family life; a summary score can be obtained by summing the three items (range 0-30, unimpaired to highly impaired). The scale's reliability and concurrent validity have been demonstrated in individuals with anxiety disorders and depression.
Time Frame: Pre-treatment, post-treatment (12 weeks after first psychotherapy session), 3-month follow-up (24 weeks after first psychotherapy appointment)
Population: OIF/OEF Veterans with PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) | Treatment as Usual (TAU)
Number analyzed (Participants) | 42 | 38
units on a scale
  Pre-Treatment | 19.0 (6.0) | 18.0 (5.1)
  Post-Treatment | 15.0 (6.7) | 16.0 (8.9)
  3-Mo Follow-Up | 15.9 (7.6) | 16.1 (8.5)

5. Secondary Outcome: Behavioral Activation Scale (BAS)
Description: The BAS is a 25-item self-report measure that assesses overall degree of behavioral activation as well as indicators of inactivation across three subscales: avoidance/rumination, work/school impairment, and social impairment. Items are rated on 7-point Likert scales (0=not at all to 6=completely). The total BAS score reflects overall level of activation with high scores reflecting higher activation (range 0 - 150).
Time Frame: Pre-treatment, post-treatment (12 weeks after 1st therapy appointment), 3-month follow-up (24 weeks after first therapy appointment)
Population: OIF/OEF Veterans with PTSD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) | Treatment as Usual (TAU)
Number analyzed (Participants) | 42 | 38
units on a scale
  Pre-Treatment | 76.0 (19.8) | 74.2 (17.7)
  Post-Treatment | 89.5 (24.4) | 82.0 (27.9)
  3-Mo Follow-Up | 79.4 (22.4) | 83.8 (27.8)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Behavioral Activation (BA) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38
Serious Adverse Events (participants affected / at risk) | 5/42 | 4/38
Other Adverse Events (participants affected / at risk) | 3/42 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation (BA) (N=42) | Treatment as Usual (TAU) (N=38)
suicidal ideation with hospitalization (Psychiatric disorders) | 2 (2) | 2 (2)
Suicidal ideation with no hospitalization (Psychiatric disorders) | 2 (2) | 2 (2)
psychotic symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
discharging firearm (Psychiatric disorders) | 0 (0) | 1 (1)
aggression with ER visit (Psychiatric disorders) | 1 (1) | 0 (0)
homicidal ideation with crisis line call (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation (BA) (N=42) | Treatment as Usual (TAU) (N=38)
very brief suicidal ideation, no hospitalization (Psychiatric disorders) | 2 (2) | 0 (0)
polymenorhea with hospitalization (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes